CLINICAL TRIAL: NCT00668837
Title: Open Label Extension to R076477-SCH-305 to Evaluate the Safety and Tolerability of Paliperidone ER in Subjects With Schizophrenia.
Brief Title: A 52 Week Open-label Extension Trial Following the Double-blind Efficacy and Safety Study R076477-SCH-305.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002944
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Paliperidone; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone

SUMMARY:
Open-Label Extension to the double-blind effectiveness and safety study R076477-SCH-305 to evaluate long-term safety and tolerability in patients with schizophrenia.

DETAILED DESCRIPTION:
The primary objective of the open-label extension trial was the long-term assessment of safety and tolerability of flexibly-dosed ER OROS paliperidone (3 to 15 mg/day) in patients with a diagnosis of schizophrenia. Other measures assessed in the extension study included: change in the total Positive and Negative Syndrome Scale (PANSS) score; change in PANSS subscale (positive and negative) scores; overall functioning, as measured by the Clinical Global Impression Scale-Severity (CGI-S); personal and social functioning, as measured by the Personal and Social Performance Scale (PSP); and quality of life parameters, as measured by the Schizophrenia Quality of Life Scale, Revision 4 (SQLS-R4). Paliperidone ER OROS® tablet formulation (3 to 15 mg/day) to be taken orally for 52 weeks

ELIGIBILITY:
Inclusion Criteria:

* Study R076477-SCH-707 enrolled patients who met the DSM-IV criteria of schizophrenia for at least 1 year
* Eligible patients were experiencing active symptoms at the time of enrollment and had a PANSS total score between 70 and 120
* The open-label extension study population comprised patients who had completed the 6-week double-blind phase of the study or who had discontinued due to lack of efficacy after at least 21 days of treatment.

Exclusion Criteria:

* Not eligible to enter the open-label phase if believed to be at significant risk for suicidal or violent behavior during the open-label extension trial
* Were pregnant
* Or had received an injection of a depot antipsychotic since entry into the preceding double-blind phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2004-02; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Flexibly-dosed ER OROS paliperidone 3 mg to 15 mg/day was safe and well tolerated in patients with schizophrenia. The safety profile was generally consistent with that observed in subjects after short-term use in the double-blind studies

SECONDARY OUTCOMES:
Findings showed stability of symptoms or further improvements in the severity of symptoms associated with schizophrenia (PANSS), personal and social functioning (PSP), global severity of illness (CGI-S), and patient-rated symptoms and well-being (SQLS)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kozma C, Dirani R, Canuso C, Mao L. Change in employment status over 52 weeks in patients with schizophrenia: an observational study. Curr Med Res Opin. 2011 Feb;27(2):327-33. doi: 10.1185/03007995.2010.541431. Epub 2010 Dec 15. PMID 21155708
- See also: A 52 week open-label extension trial following the double-blind efficacy and safety study R076477-SCH-305. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=501&filename=CR002944_CSR.pdf